CLINICAL TRIAL: NCT01536600
Title: A Multi-center, Prospective, Non-interventional Evaluation of Efficacy, Safety and Convenience of Using NovoMix 30 as Monotherapy, or in Combination With OHAs, in the Treatment of Type 2 Diabetic Patients in Routine Clinical Practice
Brief Title: Observational Study of Biphasic Insulin Aspart 30 Alone or in Combination With Oral Hypoglycaemic Agents in Subjects With Type 2 Diabetes
Acronym: PRESENT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1880
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — The insulin dose and regimen was individualised at the physician's discretion

SUMMARY:
This study is conducted in Africa, Asia and Europe. The aim of this study is to investigate biphasic insulin aspart 30 (NovoMix® 30) alone or in combination with oral hypoglycaemic agent (OHA) for type 2 diabetes management in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes whose glycaemia was not optimally controlled with current therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes who were not adequately controlled on their current therapy and who were prescribed biphasic insulin aspart 30 (NovoMix® 30)
Sampling Method: Non-Probability Sample
Enrollment: 33010 (Actual)
Dates: Start 2004-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Change in post prandial glucose (PPG)
Change in fasting glucose (FG)
Difference in prandial glucose increment (PGI)
Incidence of hypoglycaemic episodes
Adverse drug reactions (ADR)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Seoul, South Korea

REFERENCES:
- [Result] Guler S, Sharma SK, Almustafa M, Kim CH, Azar S, Danciulescu R, Shestakova M, Khutsoane D, Bech OM. Improved Glycaemic Control with Biphasic Insulin Aspart 30 in Type 2 Diabetes Patients Failing Oral Antidiabetic Drugs: PRESENT Study Results. Arch Drug Inf. 2009 Jun;2(2):23-33. doi: 10.1111/j.1753-5174.2008.00015.x. PMID 19684847
- [Result] Khutsoane D, Sharma SK, Almustafa M, Jang HC, Azar ST, Danciulescu R, Shestakova M, Ayad NM, Guler S, Bech OM; PRESENT Study Group. Biphasic insulin aspart 30 treatment improves glycaemic control in patients with type 2 diabetes in a clinical practice setting: experience from the PRESENT study. Diabetes Obes Metab. 2008 Mar;10(3):212-22. doi: 10.1111/j.1463-1326.2007.00826.x. PMID 18269636
- [Result] Shestakova M, Sharma SK, Almustafa M, Min KW, Ayad N, Azar ST, Danciulescu R, Khutsoane D, Guler S. Transferring type 2 diabetes patients with uncontrolled glycaemia from biphasic human insulin to biphasic insulin aspart 30: experiences from the PRESENT study. Curr Med Res Opin. 2007 Dec;23(12):3209-14. doi: 10.1185/030079907X253636. PMID 18005503
- [Result] Gao Y, Guo XH, Vaz JA; PRESENT Study Group. Biphasic insulin aspart 30 treatment improves glycaemic control in patients with type 2 diabetes in a clinical practice setting: Chinese PRESENT study. Diabetes Obes Metab. 2009 Jan;11(1):33-40. doi: 10.1111/j.1463-1326.2008.00904.x. Epub 2008 May 20. PMID 18494806
- [Result] Jang HC, Guler S, Shestakova M; PRESENT Study Group. When glycaemic targets can no longer be achieved with basal insulin in type 2 diabetes, can simple intensification with a modern premixed insulin help? Results from a subanalysis of the PRESENT study. Int J Clin Pract. 2008 Jul;62(7):1013-8. doi: 10.1111/j.1742-1241.2008.01792.x. Epub 2008 May 9. PMID 18479365
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com